CLINICAL TRIAL: NCT06330571
Title: The Accuracy of Clear Aligners in Maxillary Molar Distalization With and Without Attachments: A Randomized Clinical Trial.
Brief Title: The Efficiency of Clear Aligners in Maxillary Molar Distalization: A Randomized Clinical Trial.
Acronym: Aligner
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Aligners in distalization
Record Dates: First submitted 2022-03-17; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2023-07

CONDITIONS: Orthodontic Aligners
Keywords: Orthodontic, aligner, molar

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Molar distalization by aligners without attachment (Active Comparator)
  Interventions: Device: Molar distalization by aligners with attachment
- Molar distalization by aligners with attachments (Experimental)
  Interventions: Device: Molar distalization by aligners with attachment

INTERVENTIONS:
Device: Molar distalization by aligners with attachment — 1. Plaster dental models will be poured from the rubber base impression.
  2. Digital dental models will be created through scanning of plaster dental models.
  3. Planning of the aligners will be done on 3 shape clear aligner.
  4. Aligners will be fabricated on 3d printed models.
  5. Patient will receive the first aligner and will be instructed to wear it full time (except during eating and brushing) for 2 weeks.
  6. Patient will receive the following aligner after 2 weeks.
  7. Follow up visits every 4weeks until 6 months.

SUMMARY:
The aim of this study is to evaluate the accuracy of clear aligners on the amount of the maxillary molar distalization.

ELIGIBILITY:
Inclusion Criteria:

1. Age more than15 years.
2. Gender; male or female.
3. Skeletal Class I or Class II malocclusion and a bilateral half-cusp class II molar relationship that require molar distalization.
4. Mild crowding in the upper arch (≤ 4 mm).
5. Absence or previous extraction of the upper third molars.
6. Good compliance during the treatment

Exclusion Criteria:

1. Transversal dental or skeletal discrepancies.
2. Extraction treatment (except for the third molar).
3. Periodontal disease. .
4. Prosthodontics rehabilitation of the maxillary molars.

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-04-27 (Estimated); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Efficiency of aligners in molar distalization | 6 months
  T2(3shape)-T1(actual) <mm>

SECONDARY OUTCOMES:
Amount of anchorage loss | 6 months
  Linear ( mm)
Amount of molar tipping | 6 months
  Angular

CONTACTS AND LOCATIONS:
Overall Officials: Noha E Sabet, Prof, Study Chair — Ain Shams University; Marwa s Abdelatef, Phd, Study Director — Ain Shams University
Locations (1):
- Ainshams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided